CLINICAL TRIAL: NCT04271410
Title: CD19+Targeted CAR-T Cell Therapy for Relapsed/Refractory CD19+ B Cell Leukemia and Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC004
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Leukemia; Lymphoma, Large B-Cell, Diffuse; Leukemia, B-cell; Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell
Keywords: Leukemia; Lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma, Large B-Cell, Diffuse; Leukemia, B-Cell; Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CD19 CAR-T cells treat (Experimental): Patients will be be treated with CD19 CAR-T cells
  Interventions: Biological: CD19 CAR-T cells

INTERVENTIONS:
Biological: CD19 CAR-T cells — CD19 CAR-T cell therapy

SUMMARY:
This is a single arm study to evaluate the efficacy and safety of CD19-targeted CAR-T cells therapy for patients with relapsed/refractory CD19+ B Cell Leukemia and Lymphoma.

DETAILED DESCRIPTION:
There are limited options for treatment of relapse/refractory B Cell Leukemia and Lymphoma.CD19 is expressed on most B Cell Leukemia and Lymphoma cells so it is an ideal target for CAR-T. In this study, investigators will evaluate the safety and efficacy of CAR-T targeting CD19 in patients with elapsed/refractory CD19+ B Cell Leukemia and Lymphoma. The primary goal is safety and efficiency assessment, including adverse events and disease status after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent；
2. Diagnose as relapsed/refractory B Cell Leukemia and Lymphoma, and meet one of the following conditions:

   1. Failed to standard chemotherapy regimens;
   2. Relapse after complete remission, high-risk and / or refractory patients ;
   3. Relapse after hematopoietic stem cell transplantation;
3. For patients with Ph + ALL, the following conditions must be met: those who have received a standard induction chemotherapy regimen and who have not achieved complete remission after TKI treatment or have relapsed after remission (cannot tolerate TKI treatment or have contraindications to TKI treatment or the presence of TKI class) Except for drug resistant patients)；
4. Evidence for cell membrane CD19 expression；
5. All genders ，ages: 2 to 75 years；
6. The expect time of survive is above 3 months;
7. KPS>60；
8. No serious mental disorders ;
9. Left ventricular ejection fraction ≥50%
10. Sufficient hepatic function defined by ALT/AST≤3 x ULN and bilirubin≤2 x ULN;
11. Sufficient renal function defined by creatinine clearance≤2 x ULN;
12. Sufficient pulmonary function defined by indoor oxygen saturation≥92%;
13. With single or venous blood collection standards, and no other cell collection contraindications;
14. Ability and willingness to adhere to the study visit schedule and all protocol requirements.

Exclusion Criteria:

1. Previous history of other malignancy;
2. Presence of uncontrolled active infection;
3. Evidence of disorder that need the treatment by glucocorticoids;
4. Active or chronic GVHD；
5. The patients treatment by inhibitor of T cell；
6. Pregnant or breasting-feeding women;
7. Any situation that investigators regard not suitable for attending in this study (e.g. HIV , HCVinfection or intravenous drug addiction) or may affect the data analysis.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events that related to treatment | 2 years
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)
The response rate of CD19 CAR-T treatment in patients with relapse/refractory B Cell Leukemia and Lymphoma that treatment by CD19 CAR-T cells therapy | 2 years
  The response rate of CD19 CAR-T treatment will be recorded and assessed according to the National Comprehensive Cancer Network Guideline

SECONDARY OUTCOMES:
Rate of CD19 CAR-T cells in bone marrow and peripheral blood | 2 years
  In vivo (bone marrow and peripheral blood) rate of CD19 CAR-T cells were determined by means of flow cytometry
Quantity of CD19 CAR copies in bone marrow and peripheral blood | 2 years
  In vivo (bone marrow and peripheral blood) quantity of CD19 CAR copies were determined by means of qPCR
Cellular kinetics of CD19 positive cells in bone marrow | 1 years
  In vivo (bone marrow) rate and quantity of CD19 positive cells were determined by means of flow cytometry
Duration of Response (DOR) of CD19 CAR-T treatment in patients with refractory/relapsed B Cell Leukemia and Lymphoma | 2 years
  DOR will be assessed from the first assessment of CR or CRi to the first assessment of recurrence or progression of the disease or death from any cause (censored)
Progress-free survival(PFS) of CD19 CAR-T treatment in patients with refractory/relapsed B Cell Leukemia and Lymphoma | 2 years
  PFS will be assessed from the first CAR-T cell infusion to death from any cause or the first assessment of progression (censored)
Overall survival(OS) of CD19 CAR-T treatment in patients with refractory/relapsed B Cell Leukemia and Lymphoma | 2 years
  OS will be assessed from the first CAR-T cell infusion to death from any cause (censored)

CONTACTS AND LOCATIONS:
Overall Officials: Sanbin Wang, MD, Principal Investigator — 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China; Cheng Qian, PhD, Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- 920th Hospital of Joint Logistics Support Force, Kunming, Yunnan, China